CLINICAL TRIAL: NCT02274974
Title: Post-Caesarean Section Incisional Infiltration With Lidocaine Versus Lidocaine and Epinephrine;Randomized Controlled Trial.
Brief Title: Post-Caesarean Section Incisional Infiltration With Lidocaine Versus Lidocaine and Epinephrine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, AMR HELMY YEHIA, Lecturer in Obstetrics and Gynaecology, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: local infilteration of C.S
Record Dates: First submitted 2014-10-21; First posted 2014-10-27 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Pain, Postoperative
Keywords: incisional; infiltration; cs; lidocaine; epinephrine; Adverse Reaction to Topical or Infiltrative Lidocaine
MeSH Terms: conditions — Pain, Postoperative; Surgical Wound | interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lidocaine (Active Comparator): 20 ml of 2% lidocaine.
  Interventions: Drug: Lidocaine
- lidocaine and epinephrine. (Experimental): 20 ml of 2% lidocaine and epinephrine in related dose manner 1:200.000. I.e.: by adding 1/4 from ampoule of adrenaline 1mg./1ml to bottle of lidocaine Hydrochloric acid (HCL) 2% 50 ml(20mg/ml).
  Interventions: Drug: lidocaine and Epinephrine

INTERVENTIONS:
Drug: Lidocaine — •The wound of C.Swill be infiltrated before closure of the skin, with 20 ml of 2% lidocaine.
  Other Names: local anaesthetic agent.
  Arms: lidocaine
Drug: lidocaine and Epinephrine — The wound of C.S will be infiltrated before closure of the skin, with 20 ml of 2% lidocaine and epinephrine in related dose manner 1:200.000.
  Other Names: local anaesthetic agent.
  Arms: lidocaine and epinephrine.

SUMMARY:
Study to compare between efficacy of post-caesarean section infiltration with lidocaine and epinephrine versus lidocaine only to reduce post-incisional pain.

DETAILED DESCRIPTION:
assessment of adding of epinephrine to lidocaine as local infiltrator to post-caesarean section wound in prolongation of its anaesthetic effect.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing caesarean delivery under General anesthesia for various indications.
* Women refuse spinal anesthesia.

Exclusion Criteria:

* Known or suspected sensitivity to local anesthesia.
* Medical disorders induced by pregnancy (Pre-eclamptic toxemia, gestational diabetes mellitus, Hepatic diseases, homeostatic disorder)
* Medical disorders aggravated by pregnancy (cardiovascular disease, pulmonary disease, renal disease, neurological disease, metabolic or infectious diseases).
* Women who hemo-dynamically unstable.
* Lack of adequate verbal communication.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Timing of first analgesic request. | 24 hours

SECONDARY OUTCOMES:
Duration of cesarean section | 30 min to 90 min
Onset of breast breastfeeding | 24 hours
Onset of mobilization | 24 hours
  first time patient start moving after the section
Duration of hospital stay | 24 hours to 48 hours
Side effects of local infiltration of lidocaine and epinephrine | 7 days
Postoperative pyrexia | 24 hours
  <38°c

CONTACTS AND LOCATIONS:
Overall Officials: Amr H Yhia, M.D, MRCOG, Principal Investigator — Ain Shams Maternity Hospital(AinShamsMH)
Locations (1):
- Post-Caesarean Section Incisional Infiltration With Lidocaine Versus Lidocaine and Epinephrine;, Cairo, Egypt

REFERENCES:
- [Background] AbdElRhman G Ali,cairo,egypt,Post-Caerarean Section Incisional Infiltration With Lidocaine Versus Lidocaine and Epinephrine.